CLINICAL TRIAL: NCT06617572
Title: Expanded Access Protocol for Product Which Does Not Conform to the TECELRA® (Afamitresgene Autoleucel, Suspension for Intravenous Infusion) Commercial Release Specification
Brief Title: Expanded Access Protocol (EAP) for Nonconforming (NC) Afami-cel
Status: Available | Type: Expanded Access
Sponsor: USWM CT, LLC (Industry)
Responsible Party: Sponsor
Organization: USWM, LLC (dba US WorldMeds) (Industry)
Other Study IDs: ADP-0044-999
Record Dates: First submitted 2024-09-17; First posted 2024-09-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Synovial Sarcoma; Myxoid Liposarcoma
MeSH Terms: conditions — Sarcoma, Synovial; Liposarcoma, Myxoid

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Genetic: Non-conforming afamitresgene autoleucel — Non-conforming afamitresgene autoleucel, suspension for intravenous infusion (NC afami-cel), single dose administration

SUMMARY:
The purpose of this expanded access protocol (EAP) is to provide controlled access to Afamitresgene autoleucel, suspension for intravenous infusion that does not meet the commercial release specification (NC afami-cel). This EAP will be conducted at authorized treatment centers where TECELRA® is being administered and where the EAP is approved to be conducted. Patients who are prescribed TECELRA® , sign the informed consent form, and meet all entry criteria will be eligible to participate in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient must provide written informed consent prior to participating in this protocol
* Patient must have been prescribed TECELRA®
* Patient's commercially manufactured product does not meet the commercial release specification
* Repeat manufacture is not feasible or is not clinically appropriate per Investigator assessment in consultation with Adaptimmune
* Repeat leukapheresis is not feasible or is not clinically appropriate per Investigator assessment
* The Investigator has confirmed a favorable benefit:risk profile, following sponsor evaluation of the NC afami-cel, and deems proceeding with treatment under this EAP is in the best interest of the patient
* Patient deemed medically fit and stable to receive NC afami-cel per Investigator assessment
* Female patients with reproductive potential must have a negative serum or urine pregnancy test within 7 days of initiating lymphodepleting chemotherapy

Exclusion Criteria:

* Patient has contraindication(s) as per the TECELRA® USPI
* Do not use TECELRA® in adults who are heterozygous or homozygous for HLA-A*02:05P

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Mayo Arizona, Phoenix, Arizona
  - Stanford Hospital and Clinics, Stanford, California
  - Mayo Florida, Jacksonville, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Centre, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas